CLINICAL TRIAL: NCT03702725
Title: A Phase I Study of Ibrutinib (PCI-32765) in Combination With Revlimid/Dexamethasone (Rd) in Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Ibrutinib in Combination With Revlimid/Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-15
Record Dates: First submitted 2018-08-31; First posted 2018-10-11 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Refractory Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Refractory Multiple Myeloma; Ibrutinib
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — ibrutinib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will consist of three different drug levels of Ibrutinib, Lenalidomide, and Dexamethasone.
  Dose Escalation (Ibrutinib, Lenalidomide, Dexamethasone Combination)
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Dexamethasone
- Dose Expansion (Experimental): Dosage of the combination will depend on the determine of maximum tolerated dose learned from the Dose Escalation phase.
  Dose Expansion (Ibrutinib, Lenalidomide, Dexamethasone Combination)
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib administered on every day of each 28 day cycle. Dosage depends on timing of patient enrollment and dosage tolerance by patients already enrolled.
  Other Names: Imbruvica
Drug: Lenalidomide — Lenalidomide administered on days 1-21 of each 28 day cycle. Dosage depends on findings from Dose Escalation phase.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone administered on days 1, 8, 15, and 22 of every 28 day cycle. Dosage depends on findings from Dose Escalation phase.
  Other Names: Decadron

SUMMARY:
This is a registration, open-label phase 1 study of the combination of ibrutinib/lenalidomide:/dexamethasone in women and men with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
The study will be completed in two parts: Dose escalation and dose expansion.

Dose Escalation Starting doses of ibrutinib and lenalidomide will be assigned at the time of registration. A minimum of 2 or a maximum of 6 patients will be accrued to a given dose level. Doses will not be escalated in any individual patient.

If none of the first 3 patients treated at a given dose level develops a dose limiting toxicity during the first cycle of treatment, enrollment to the dose level will be closed and enrollment will reopen at next higher dose level. If there are no other higher dose levels to be tested, three additional patients will be enrolled at the current dose level to confirm maximum tolerated dose. If one of the first 3 patients treated at a given dose level develops a dose limiting toxicity during the first cycle of treatment, three additional patients will be enrolled onto the current dose level. If, at any time in the enrollment of these 3 additional patients, a patient develops a dose limiting toxicity, enrollment will be closed to this dose level. Enrollment will be re-opened to the next lower dose level if fewer than 6 patients have been treated at that dose level. If none of these 3 additional patients develops a dose limiting toxicity during the first cycle of treatment, enrollment to this dose level will be closed and enrollment will reopen at next higher dose level. If there are no other higher dose levels to be tested, this will be considered the maximum tolerated dose.

Patients will return to the clinic every 28 days for physical exams, laboratory assessments and review of side effects.

Patients who do not have disease progression and have not experienced unacceptable toxicities will be eligible to continue protocol treatment at their current dose level until disease progression, unacceptable toxicity, or refusal. Those patients who have not experienced progression of disease but have unacceptable toxicity may be eligible for re-treatment at a lower dose.

Part 2: Dose Expansion Once the maximum tolerated dose has been established or determined, 4-10 additional patients will be treated at the maximum tolerated dose of lenalidomide and ibrutinib at the same schedule as above. Dexamethasone will be given at the same dose as in the dose escalation portion of the study.

Patients who discontinue treatment for protocol defined reasons will go to survival follow-up. Once a patient has entered the survival follow-up phase of the trial, his/her therapy is at the discretion of the treating physician. Patients' charts will be reviewed for progression and survival endpoints during visits with treating physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Appendix I).
3. Symptomatic multiple myeloma (MM) (as defined by revised IMWG criteria) with measurable disease, defined here as having at least one of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL
   * ≥200 mg of monoclonal protein in the urine on 24 hour electrophoresis
   * Serum immunoglobulin free light chain (FLC): involved FLC ≥ 10 mg/dL (≥ 100 mg/L) AND abnormal serum immunoglobulin kappa to lambda free light chain ratio.
4. At least 1 prior therapy with demonstrated disease progression following the most recent line of treatment.
5. Progression of disease within 60 days of completion of last therapeutic regimen or the failure to achieve minimal response while on last treatment (according to IMWG).

   • Patients should not have progressed on lenalidomide at a dose of more than 10mg
6. No prior treatment with ibrutinib or any other protein kinase inhibitory drug or drug targeting the b-cell receptor (BCR) signal transduction pathway.
7. Patients with prior daratumumab and allogeneic stem cell transplant are included.
8. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN, except if on anticoagulation for medical reasons in which case INR should be ≤ 3
9. Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to registration, with the exception of pegylated G-CSF (pegfilgrastim) and darbopoeitin which require at least 14 days prior to screen and enrollment defined as:

   * Absolute neutrophil count (ANC) ≥1000/mm3 independent of growth factor support.
   * Transfusion independent platelet counts ≥75,000/mm3 (or ≥50,000/mm3 if bone marrow involvement is ≥50%).
   * Hemoglobin level ≥ 8 g/dL, independent of transfusion support.
10. Biochemical values must be within the following limits within 7 days prior to registration

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN).
    * Total bilirubin ≤ 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
    * Serum creatinine ≤ 2 x ULN or GFR > 30 ml/min based on either the estimated Glomerular Filtration Rate (Crockcoft Gault) or measured GFR from 24-hour urine sample. Study participants with GFR 30-50 ml/min will be treated according to manufacturer's instruction with lenalidomide 10mg rather than 25 mg.
11. Ability to understand and willingness to sign a written informed consent form (ICF).
12. Ability to adhere with the study visit schedule and other protocol procedures.
13. A negative pregnancy test will be required for all women of child bearing potential within 7 days prior to registration. Breast feeding is not permitted.
14. Fertility requirements

    * Female patients with child bearing potential must have a negative pregnancy test at least 7 days before starting treatment drugs.
    * Male subject must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.
    * Female patients must be either post-menopausal, free from menses ≥ 2yrs, surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from sexual activity starting from screening and for 90 days after lenalidomide treatment
    * Female patients of childbearing potential must agree to comply with the fertility and pregnancy test requirements dictated by the Rev-Assist program.
15. Willingness to provide blood and tissue samples for correlative research purposes

Exclusion Criteria:

1. Prior history of: Polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes (POEMS) syndrome, osteosclerotic myeloma, Crow-Fukase syndrome, primary amyloidosis or plasma cell leukemia.
2. Radiotherapy within 21 days of registration. However, if the radiation portal was localized to single lesion or fracture site and covered by ≤ 5% of the bone marrow reserve (by investigator estimate), the subject may be enrolled irrespective of the end date of radiotherapy.
3. Prior chemotherapy:

   * Alkylators (e.g. melphalan, cyclophosphamide) ≤ 21 days prior to registration and/or monoclonal antibody ≤ 6 weeks prior to first administration of study treatment.
   * Anthracyclines ≤ 21 days prior to registration.
   * High dose corticosteroids, immune modulatory drugs (thalidomide or lenalidomide), or proteasome inhibitors (bortezomib or carfilzomib) ≤ 14 days prior to registration.
4. No concomitant high dose corticosteroids (concurrent use of corticosteroids). EXCEPTION: Patients may be on chronic steroids (maximum dose 10 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, i.e., adrenal insufficiency, rheumatoid arthritis, etc.
5. Currently active, clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to registration or baseline QTcF of > 470.
6. Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
7. History of prior malignancy, with the exception of the following:

   * Malignancy treated with curative intent and with no known active disease present for more than 3 years prior to registration and felt to be at low risk for recurrence by treating physician;
   * Adequately treated non melanoma skin cancer or lentigo maligna without current evidence of disease; or
   * Adequately treated breast or cervical carcinoma in situ without current evidence of disease.
8. Peripheral neuropathy Grade > 2 on clinical examination within 14 days prior to registration.
9. Uncontrolled diabetes mellitus.
10. Currently active systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
11. Use of antibiotics for treatment of infection within 14 days prior to registration
12. Recent infection requiring systemic treatment that was completed within 14 days of registration.
13. Known infection with human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) or any uncontrolled active systemic infection.

    Note: Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result within 14 days prior to registration.
14. History of stroke or intracranial hemorrhage within 6 months prior to registration.
15. Patients who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or patient who requires continuous treatment with a strong CYP3A inhibitor (Appendix II).
16. Currently active, clinically significant hepatic impairment (Child-Pugh class B or C) according to the Child Pugh classification (Appendix III).
17. Lactating or pregnant
18. Major surgery within 4 weeks prior to registration
19. Known bleeding disorders (e.g. von Willebrand's disease or hemophilia).
20. Allergies and adverse drug reactions: history of allergy to study drug components
21. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
22. Any life-threatening illness, medical condition, or organ systemic dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
23. Unresolved toxicities from prior anti-cancer therapy, defined as not having resolved to CTCAE Version 5.0, Grade 0 or 1, with the exception of alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Yvonne A. Efebera, MD, Study Chair — Ohio State University Comprehensive Cancer Center; Jacob P. Laubach, MD, Study Chair — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Loyola University Medical Center, Maywood, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center/James Cancer Hospital, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Richardson P, Jagannath S, Hussein M, Berenson J, Singhal S, Irwin D, Williams SF, Bensinger W, Badros AZ, Vescio R, Kenvin L, Yu Z, Olesnyckyj M, Zeldis J, Knight R, Anderson KC. Safety and efficacy of single-agent lenalidomide in patients with relapsed and refractory multiple myeloma. Blood. 2009 Jul 23;114(4):772-8. doi: 10.1182/blood-2008-12-196238. Epub 2009 May 26. PMID 19471019
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Murray MY, Zaitseva L, Auger MJ, Craig JI, MacEwan DJ, Rushworth SA, Bowles KM. Ibrutinib inhibits BTK-driven NF-kappaB p65 activity to overcome bortezomib-resistance in multiple myeloma. Cell Cycle. 2015;14(14):2367-75. doi: 10.1080/15384101.2014.998067. Epub 2015 Jan 7. PMID 25565020
- [Background] Yang Y, Shi J, Gu Z, Salama ME, Das S, Wendlandt E, Xu H, Huang J, Tao Y, Hao M, Franqui R, Levasseur D, Janz S, Tricot G, Zhan F. Bruton tyrosine kinase is a therapeutic target in stem-like cells from multiple myeloma. Cancer Res. 2015 Feb 1;75(3):594-604. doi: 10.1158/0008-5472.CAN-14-2362. Epub 2015 Jan 14. PMID 25589346
- [Background] Bam R, Ling W, Khan S, Pennisi A, Venkateshaiah SU, Li X, van Rhee F, Usmani S, Barlogie B, Shaughnessy J, Epstein J, Yaccoby S. Role of Bruton's tyrosine kinase in myeloma cell migration and induction of bone disease. Am J Hematol. 2013 Jun;88(6):463-71. doi: 10.1002/ajh.23433. Epub 2013 Mar 28. PMID 23456977
- [Background] Rushworth SA, Bowles KM, Barrera LN, Murray MY, Zaitseva L, MacEwan DJ. BTK inhibitor ibrutinib is cytotoxic to myeloma and potently enhances bortezomib and lenalidomide activities through NF-kappaB. Cell Signal. 2013 Jan;25(1):106-12. doi: 10.1016/j.cellsig.2012.09.008. Epub 2012 Sep 11. PMID 22975686
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Yang Y, Shaffer AL 3rd, Emre NC, Ceribelli M, Zhang M, Wright G, Xiao W, Powell J, Platig J, Kohlhammer H, Young RM, Zhao H, Yang Y, Xu W, Buggy JJ, Balasubramanian S, Mathews LA, Shinn P, Guha R, Ferrer M, Thomas C, Waldmann TA, Staudt LM. Exploiting synthetic lethality for the therapy of ABC diffuse large B cell lymphoma. Cancer Cell. 2012 Jun 12;21(6):723-37. doi: 10.1016/j.ccr.2012.05.024. PMID 22698399
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Bishop GA, Haxhinasto SA, Stunz LL, Hostager BS. Antigen-specific B-lymphocyte activation. Crit Rev Immunol. 2003;23(3):149-97. doi: 10.1615/critrevimmunol.v23.i3.10. PMID 14584878
- [Background] Chang BY, Francesco M, De Rooij MF, Magadala P, Steggerda SM, Huang MM, Kuil A, Herman SE, Chang S, Pals ST, Wilson W, Wiestner A, Spaargaren M, Buggy JJ, Elias L. Egress of CD19(+)CD5(+) cells into peripheral blood following treatment with the Bruton tyrosine kinase inhibitor ibrutinib in mantle cell lymphoma patients. Blood. 2013 Oct 3;122(14):2412-24. doi: 10.1182/blood-2013-02-482125. Epub 2013 Aug 12. PMID 23940282
- [Background] Herman SE, Gordon AL, Hertlein E, Ramanunni A, Zhang X, Jaglowski S, Flynn J, Jones J, Blum KA, Buggy JJ, Hamdy A, Johnson AJ, Byrd JC. Bruton tyrosine kinase represents a promising therapeutic target for treatment of chronic lymphocytic leukemia and is effectively targeted by PCI-32765. Blood. 2011 Jun 9;117(23):6287-96. doi: 10.1182/blood-2011-01-328484. Epub 2011 Mar 21. PMID 21422473
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Rajkumar SV, Jacobus S, Callander NS, Fonseca R, Vesole DH, Williams ME, Abonour R, Siegel DS, Katz M, Greipp PR; Eastern Cooperative Oncology Group. Lenalidomide plus high-dose dexamethasone versus lenalidomide plus low-dose dexamethasone as initial therapy for newly diagnosed multiple myeloma: an open-label randomised controlled trial. Lancet Oncol. 2010 Jan;11(1):29-37. doi: 10.1016/S1470-2045(09)70284-0. Epub 2009 Oct 21. PMID 19853510
- [Background] Geiss GK, Bumgarner RE, Birditt B, Dahl T, Dowidar N, Dunaway DL, Fell HP, Ferree S, George RD, Grogan T, James JJ, Maysuria M, Mitton JD, Oliveri P, Osborn JL, Peng T, Ratcliffe AL, Webster PJ, Davidson EH, Hood L, Dimitrov K. Direct multiplexed measurement of gene expression with color-coded probe pairs. Nat Biotechnol. 2008 Mar;26(3):317-25. doi: 10.1038/nbt1385. Epub 2008 Feb 17. PMID 18278033

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Starting DL): Ibrutinib 560 mg on Days 1-28,> Lenalidomide 15 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22>
  > Every 28 days
- Dose Level 2: Ibrutinib 560 mg on Days 1-28,> Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22>
  > Every 28 days
- Dose Level 3: Ibrutinib 840 mg on Days 1-28,> Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22>
  > Every 28 days
Period: Overall Study
Arm/Group | Dose Level 1 (Starting DL) | Dose Level 2 | Dose Level 3
Started | 6 | 3 | 4
Completed | 6 | 3 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (Starting DL) | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 6 | 3 | 4 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [52 to 64] | 68 [61 to 73] | 64.5 [63.5 to 68] | 64 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 8
  Male | 3 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 3 | 11
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 5 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: DLTs were grade 4 thrombocytopenia; grade 4 neutropenia lasting > 5 days or febrile neutropenia; grade 3 thrombocytopenia with bleeding or platelet transfusion; grade 3-4 hyperglycemia or a thrombotic/embolic event; or grade 3-4 non-hematologic toxicity (except grade 3 nausea, diarrhea, and vomiting), that were at least probably related to treatment, treatment delays ≥ 21 days for toxicity, and treatment-related death.
Time Frame: During cycle 1 (28-day cycle)
Population: Eligible patients who started protocol treatment were excluded from the determination of MTD if they failed to completed one cycle of treatments for reasons other than toxicity. Specifically. two patient assigned to DL3 were excluded from MTD determination: one developed COVID-19 infection and the other received 280 mg/day of IBR instead of the assigned 840 mg/day dose during cycle 1.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 (Starting DL): Ibrutinib 560 mg on Days 1-28,
  > Lenalidomide 15 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  >
  > Every 28 days
- Dose Level 2: Ibrutinib 560 mg on Days 1-28,
  > Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  >
  > Every 28 days
- Dose Level 3: Ibrutinib 840 mg on Days 1-28,
  > Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  >
  > Every 28 days
Arm/Group | Dose Level 1 (Starting DL) | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 3 | 2
Participants | 1 | 0 | 0
Statistical Analysis 1: Comparison: Dose Level 1 (Starting DL) vs Dose Level 2 vs Dose Level 3; Test type: Other; Estimate value DL 3

2. Primary Outcome: Maximum Toxicity Grade
Description: The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity as well as the percentage of patients developing a severe degree (Grade 3 or higher) will be determined. Adverse Events were graded using CTCAE v4.0.
Time Frame: Up to 34 month
Population: All eligible patients who began protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 Starting Cohort: Ibrutinib 560 mg on Days 1-28,
  > Lenalidomide 15 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  >
  > Every 28 days
Arm/Group | Dose Level 1 Starting Cohort | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 3 | 4
Participants
  Grade 3 | 4 | 3 | 3
  Grade 4 | 1 | 0 | 1
  Grade 5 | 1 | 0 | 1

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival time is the time from study entry to the documentation of disease progression or death due to any cause.
Time Frame: 34 Months
Population: Per-protocol - all eligible patients who initiated protocol treatment regardless of DL received
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Dose Level 1 Starting Cohort: Ibrutinib 560 mg on Days 1-28,
  * Lenalidomide 15 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  * Every 28 days
- Dose Level 2: Ibrutinib 560 mg on Days 1-28,
  * Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  * Every 28 days
- Dose Level 3: Ibrutinib 840 mg on Days 1-28,
  * Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  * Every 28 days
Arm/Group | Dose Level 1 Starting Cohort | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 3 | 4
days | 215 [56 to NA] — There are not enough events to calculate upper confidence bound. | 106 [85 to NA] — There are not enough events to calculate upper confidence bound. | 102 [56 to NA] — There are not enough events to calculate upper confidence bound.

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as time from registration to death due to any cause.
Time Frame: 34 Months
Population: Per-protocol - all eligible patients who initiated protocol treatment regardless of DL received
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dose Level 1 Starting Cohort | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 3 | 4
Days | NA [NA to NA] — median and confidence interval not estimable due to an insufficient number of participants with events | 404 [208 to NA] — median and confidence interval not estimable due to an insufficient number of participants with events | 254 [80 to NA] — median and confidence interval not estimable due to an insufficient number of participants with events

5. Secondary Outcome: Duration of Response
Description: The duration of response is the time from initiation of first response to first documentation of disease progression or death. Patients who have not progressed will be censored at the date of their last disease evaluation.
Time Frame: 34 Months
Population: All eligible patients who met IMWG criteria for CR, VGPR, or PR on two consecutive evaluations at least 4 weeks apart
Measure: Number; unit: months
Arm/Group | Dose Level 1 (Starting DL) | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 1 | 0 | 1
months | 7.1 |  | 3.1

6. Secondary Outcome: Objective Response Rate
Description: The objective response rate is the percent of patients who meet the International Myeloma Working Group Response Criteria for sCR, CR, VGPR, or PR on two consecutive evaluations at least 4 weeks apart among the patients who began study treatment. A 90% binomial confidence interval will be constructed for the overall objective response rate.
Time Frame: Up to 34 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Dose Level 2: * Lenalidomide 15 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  * Every 28 days Ibrutinib 560 mg on Days 1-28,
  * Lenalidomide 25 mg on Days 1-21 Dexamethasone 40 mg on Days 1,8,15, 22
  * Every 28 days
Arm/Group | Dose Level 1 Starting Cohort | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 3 | 4
percentage of participants | 16.7 [0.9 to 58.2] | 0 [0 to 63.2] | 25 [1.3 to 75.1]

ADVERSE EVENTS:
Time Frame: Up to 34 months
Arm/Group | Dose Level 1 (Starting DL) | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/3 | 3/4
Serious Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 4/4
Other Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Starting DL) (N=6) | Dose Level 2 (N=3) | Dose Level 3 (N=4)
Anemia (Blood and lymphatic system disorders) | 4 (8) | 3 (6) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 3 (9) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (5) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (9) | 3 (6) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 2 (6) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (7) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (2) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (5) | 2 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (3) | 2 (4) | 3 (5)
Weight loss (Investigations) | 1 (1) | 2 (3) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 3 (8) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Starting DL) (N=6) | Dose Level 2 (N=3) | Dose Level 3 (N=4)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT03702725/Prot_SAP_000.pdf